CLINICAL TRIAL: NCT03773770
Title: Expanded Access to Triheptanoin
Status: Available | Type: Expanded Access
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX007-EAP
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Long Chain Fatty Acid Oxidation Disorders
Keywords: Expanded Access; Compassionate Use; Carnitine Palmitoyltransferase Deficiency; CPT I; CPT II; Very Long Chain acyl-CoA Dehydrogenase Deficiency; VLCAD; Long Chain 3-hydroxy-acyl-CoA Dehydrogenase Deficiency; LHCAD; Trifunctional Protein Deficiency; TFP; Carnitine-acylcarnitine Translocase Deficiency; CACT; LC-FAOD
MeSH Terms: conditions — VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Carnitine-Acylcarnitine Translocase Deficiency | interventions — triheptanoin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Triheptanoin — Liquid for oral (PO) or enteral tube administration
  Other Names: UX007

SUMMARY:
Expanded access may be provided for qualified patients who have limited treatment options and are not eligible for a clinical trial.

DETAILED DESCRIPTION:
Long Chain Fatty Acid Oxidation Disorders (LC-FAOD) and other Non-FAOD conditions, where applicable: Expanded access may be available outside of the US in countries prior to approval by the local regulatory agencies.

For full details, please visit the links provided below.

ELIGIBILITY:
- The participant must not be eligible for a UX007 clinical trial

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc

REFERENCES:
- See also: Access to Investigational Therapies / Requesting Access — https://www.ultragenyx.com/our-purpose/supporting-access-for-patients/?#investigational-therapies
- See also: Dojolvi Patient and Prescribing Information Page — https://www.dojolvi.com/